CLINICAL TRIAL: NCT01174186
Title: Intestinal Inflammation in Ankylosing Spondylitis Assessed by Fecal Calprotectin, Capsular Endoscopy and Colonoscopy and the Effects of Adalimumab on Mucosal Healing
Brief Title: Intestinal Inflammation in Ankylosing Spondylitis and the Effects of Adalimumab on Mucosal Healing
Acronym: INTASAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Collaborators: Abbott (Industry); Medtronic - MITG (Industry); Central Denmark Region (Other)
Responsible Party: Principal Investigator, Rene Oestgaard, René Østgård, MD, Regional Hospital Denmark, medical department, Regionshospitalet Silkeborg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4682724
Record Dates: First submitted 2010-07-16; First posted 2010-08-03 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Spondyloarthritis; Enterocolitis
MeSH Terms: conditions — Spondylarthritis; Enterocolitis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spondyloarthritis and calprotectin elevated (Active Comparator): Spondylitis patients with elevated levels of fecal calprotectin. Patients are treated with adalimumab
  Interventions: Drug: Adalimumab
- Spondyloarthritis and calprotectin normal (Active Comparator): Spondylitis patients with normal levels of fecal calprotectin. Patients are treated with adalimumab.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Tumor Necrosis Factor (TNF) alpha inhibitor given 40 mg subcutaneously every other week except the first time where 80 mg is given
  Other Names: Humira

SUMMARY:
Studies with intestinally asymptomatic patients with spondyloarthritis showed that approximately 1/3 had visible ulcers in the colon by scopic examinations and 2/3 had changes detectable by microscopy. Only those patients who improved in arthritis symptoms showed improvement in colonic changes. In these studies only colon and the terminal ileum was examined. Inflammation of the small intestine was not examined. Newer studies have shown an immunological link between Crohns disease and spondyloarthritis but not ulcerative colitis. The investigators wish to examine the small intestine in these patients before and after treatment, since they expect to find ulcers there linking spondyloarthritis to Crohns disease and healing after treatment.

DETAILED DESCRIPTION:
Patients with inflammatory axial spondyloarthritis according to the assessment group in ankylosing spondylitis (ASAS) criteria (8) and active disease assessed by a physician are recruited in the outpatient clinics of the rheumatology departments, provided that the patient under normal circumstances is expected to benefit from TNF-alpha inhibitor treatment and full fill the criteria for treatment. Screening with a view to participating in the study is carried out in accordance with the inclusion and exclusion criteria. Oral and written patient information about the study, the patient's signing of the informed consent form and the signing of the patient's power of attorney in accordance with the study protocol are also a condition for the inclusion. The including physician will ensure that a potential participant is informed about the right to at least 1 hour's reflection time and the right to have a friend/family member present at the information interview.

If the patient meets the basis for the participation in the study the informed consent form and the power of attorney are signed.

The screened patients are not coded but are identified using their Civil Registration Number (CPR) for several reasons. The study is open-label, which removes the need for blinding of patients as well as investigator. Blood samples are booked electronically and printed labels with CPR number are put on the test tubes for both immediate analysis and storage. This guarantees a more fail-safe method for handling of various analyses, since this procedure is similar to the routine procedure. We find this to be the safest system as the method, by which labels with CPR number follow the patient has been thoroughly tested.

Source data will be kept in the Danish Biologics Online Registry (DANBIO registry) for clinical measures, the electronic patient file for lab data and the paper file for imaging data. Data validity and completeness is controlled by external "good clinical practice" monitoring.

Adalimumab will be supplied as a sterile solution without preservatives for subcutaneous injection in 1 ml prefilled syringes containing adalimumab 40 mg/0.8 ml, to be self-injected by the patient every 2 weeks until week 20. After week 20 patients continue adalimumab treatment 40 mg every other week but may change to injections with pens containing the same drug and dosage. The drug is injected under the skin of the abdomen or the thigh. All patients will be instructed by the study personnel in correct sterile subcutaneous injection of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18 years and ≤45 years) with axial SpA according to the ASAS criteria
* Active SpA assessed by physician.
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4.
* Faecal calprotectin ≥ 100mg/kg.
* Negative pregnancy test (serum-HCG) for women of childbearing age before the start of the study. (Women not of childbearing age are defined as postmenopausal for at least 1 year or surgically sterilised (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)). Women of childbearing age included in the study will be required to use contraception during the entire study period (i.e. one of the following: contraceptive pills, intrauterine device, depot injection of gestagen, subdermal implant, hormonal vaginal ring or transdermal patch). In addition, contraception must be used following any discontinuation of the study drug for a period of 150 days.
* Ability and willingness to self-administer the subcutaneous injections or have a person available to administer the injections.
* Ability and willingness to give written informed consent and meet the requirements of the study protocol.

Exclusion Criteria:

* Diagnosed inflammatory bowel disease or high risk of intestinal stricture (previous abdominal stricture, radiation of abdomen, major abdominal surgery).
* Non steroid anti inflammatory Drugs (NSAID) ingestion less than 4 weeks before inclusion.
* Psoriasis
* Persons with latent Tuberculosis (TB)(positive Mantoux skin test (>10 mm), positive cultivation for mycobacteria in tissue samples and/or chest X-ray indicating TB) or other risk factors for activation of untreated latent TB.
* Current or recurrent infections or serious infections requiring hospitalisation or treatment with intravenous antibiotics within the last 30 days or oral antibiotics within the last 14 days before inclusion.
* Positive serology for Hepatitis B or C indicating active infection.
* Medical history of positive HIV status (in case of suspicion control of HIV test).
* Medical history of histoplasmosis or listeriosis.
* Previous cancer or lymphoid proliferative disease except completely well-treated cutaneous squamous cell carcinoma, basal cell carcinoma or cervical dysplasia.
* Previous diagnosis or signs of demyelinising diseases of the central nervous system (e.g. optic neuritis, disturbance of vision, disturbed gait/ataxia, facial paresis, apraxia).
* Severe renal insufficiency (creatinine clearance < 35 ml/min - normogram).Affected hepatic function: Liver enzymes > 3 x above the normal limit.
* Clinically significant drug or alcohol abuse in the last year or daily current alcohol consumption.
* Diabetes, unstable ischemic heart disease, heart failure (NYHA III-IV), recent apoplexia cerebri (within 3 months), chronic leg ulcer and any other condition (e.g. indwelling catheter) which at the discretion of the investigator means that participation in the protocol would entail a risk for the person in question.
* Anticoagulant treatment.
* Pregnancy or breast-feeding.
* Other clinically significant inflammatory rheumatologic diseases that cannot be related to spondyloarthritis
* Current parvovirus B 19 infection.
* Glucocorticosteroid treatment within the last 4 weeks (except nasal and inhalation steroids).
* Contraindication to study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Glerup, M.D., Study Chair — Regional Hospital Silkeborg, medical department; René D Oestgaard, M.D., Study Director — Regional Hospital Silkeborg, medical department; Bent Deleuran, M.D., Principal Investigator — Department of Medical Microbiology and Immunology Aarhus University
Locations (4):
- Denmark (4):
  - Department of Rheumatology U, Aarhus Hospital, Aarhus
  - Regional Hospital of Horsens, Department of Medicine, Horsens
  - Regional Hospital of Randers, Department of Medicine, Randers
  - Regional Hospital of Silkeborg, Silkeborg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SpA patients eligible for anti-TNF treatment as described by ASAS guidelines were included from outpatient clinics in Northern Jutland, Denmark. Patients were included over a 2 years and three months time span
Pre-assignment Details: Patient on current non-steroidal anti-inflammatory (NSAID) treatment were subjected to a 4 week long wash-out period, because NSAID can cause falsely elevated fecal calprotectin levels
Groups:
- Calprotetin Elevated: Spondylitis patients with active inflammation and elevated calprotectin
  Adalimumab: Tumor Necrosis Factor (TNF) alpha inhibitor given 40 mg subcutaneously every other week except the first time where 80 mg is given
- Calprotectin Normal: Spondylitis patients with active inflammation and normal calprotectin
  Adalimumab: Tumor Necrosis Factor (TNF) alpha inhibitor given 40 mg subcutaneously every other week
Period: Overall Study
Arm/Group | Calprotetin Elevated | Calprotectin Normal
Started | 15 (Patients were included over three years) | 15
Completed | 15 | 12
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: n=15 in each group was determined by power calculations from previous pilot trials on differences in calprotectin
Groups:
- Total: Total of all reporting groups
Arm/Group | Calprotetin Elevated | Calprotectin Normal | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  Denmark | 15 | 15 | 30
Bath Ankylosing Spondylitis Disease Activity Index >4 [Number; unit: participants] — Patient answered composite index for describing disease activity. Range from 0-10. Higher scores indicate higher disease activity
  participants | 15 | 15 | 30
No effect of NSAID [Number; unit: participants] | 15 | 15 | 30
Expert opinion of active disease [Number; unit: participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change Lewis Score Index
Description: Lewis' score describes the amount of inflammation seen optically by capsular endoscopy.
  Gralnek et al. devised and validated the Lewis score index, based on three endoscopic parameters: villous edema, ulcer and stenosis/stricture. Using these parameters, the authors established a score range of 8-4,800 points where: LS < 135 reflects normal mucosal appearances, LS 135-790 mild mucosal inflammatory change and an LS value ≥790 moderate to severe mucosal inflammatory changes.
  The patients had endoscopy performed at baseline and again after 20 weeks. The number of patients improving was compared to number of patients deteriorating
Time Frame: 20 weeks
Population: Because endoscopy has a small risk for perforation. The study was designed so only patients with active inflammation at baseline had follow-up endoscopy performed. Because all patients with normal calprotectin levels had normal endoscopy, follow-up was only performed on this group of patients.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Calprotetin Elevated
Number analyzed (Participants) | 15
units on a scale | -225 [-493 to -112]

2. Primary Outcome: Change in Intestinal Inflammation Measured by Faecal Calprotectin
Description: Feacal calprotectin is a protein and a marker of the degree of inflammation in the intestine, but not the site of inflammation.
  We measured the level calprotectin continuously in each of the patients. Difference was inferred by repeated measurement ANOVA
Time Frame: Baseline to 52 weeks
Population: 15 patients in each group was included. 3 in the calprotectin negative group patients did not fulfill the entire study period (1 lost to follow-up, 2 withdrew consent).
  Data analysed as last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | Calprotetin Elevated | Calprotectin Normal
Number analyzed (Participants) | 15 | 15
mg/g | 44 [30 to 147] | 30 [30 to 30]

3. Secondary Outcome: Spondyloarthritis Consortium of Canada Score
Description: Inflammation on MRI assessed by the Spondyloarthritis Consortium of Canada score and a Danish scoring method
Time Frame: one year
Reporting Status: Not Posted

4. Secondary Outcome: Assessment Group in Ankylosing Spondylitis (ASAS) Core Set for Clinical Practice
Description: clinical measurements of inflammation in spondyloarthritis patients as described by the Assessment Group in Ankylosing Spondylitis (ASAS)
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire follow-up period of one year
Arm/Group | Calprotetin Elevated | Calprotectin Normal
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calprotetin Elevated (N=15) | Calprotectin Normal (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient admitted with abdominal pains after consuming alcohol. Was discharged the next day after lab results came out normal and abdominal pains had subsided
Gastro intestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Admitted to hospital because of severe anemia. Patient was bleeding from a Meckel's diverticulum

LIMITATIONS AND CAVEATS:
15 participants in each group is not many, but the number was selected based on an a priori analysis.

NSAID wash-out period of 4 weeks was chosen as best estimate. Loading dose of adalimumab was given to calprotectin elevated group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No